CLINICAL TRIAL: NCT06329193
Title: Effects of Mid-Season Camp Period Loading on Sports Injury Anxiety and Physical Performance of Professional Male Soccer Players
Brief Title: Effects of Mid-Season Camp Period Loading on Sports Injury Anxiety and Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Erhan Seçer, Lecturer, Celal Bayar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CBU-FTR-ES-O4
Record Dates: First submitted 2024-03-19; First posted 2024-03-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Exercise; Athletic Performance
MeSH Terms: conditions — Anxiety Disorders; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Group (Experimental): The 3-week mid-season camp period loading at sea level, including daily gym and field-based exercise interventions, five days a week, will be applied to the participants in the sports club's gym and soccer field.
  Interventions: Other: Mid-Season Camp Period Loading

INTERVENTIONS:
Other: Mid-Season Camp Period Loading — The daily gym included warm-up protocol (dynamic stretching of the major muscle groups of the upper and lower extremities and jogging), crunches, sit-ups, reverse sit-ups, prone bridge, side bridge, bench press, mini squat (with body weight and/or ancillary equipment), lunge (with body weight and/or ancillary equipment), leg extension, leg curl, leg press, calf raises (with body weight and/or ancillary equipment), and cool-down protocol (dynamic stretching of the major muscle groups of the upper and lower extremities). The field-based exercises included warm-up protocol (dynamic stretching of the major muscle groups of the upper and lower extremities and jogging), dynamic balance (with different balance trainer such as Both Sides Utilized [BOSU], trampoline), tactical training, passing, dribbling, and shooting practice, agility and speed practice, and cool-down protocol (dynamic stretching of the major muscle groups of the upper and lower extremities)

SUMMARY:
The aim of this study is to investigate the effects of 3-week mid-season camp period loading on sports injury anxiety level and physical performances of professional male soccer players.

DETAILED DESCRIPTION:
According to the periodization theory, the seasonal training process of soccer players is divided into four periods such as pre-season, early competition, late competition, and transition. In general, these periods aim to prepare soccer players for the competitive season, improve their fitness and physical performance, and reduce the risk of sports injuries. Therefore, the loading applied to soccer players during these camp periods are the key determinants of physical performance enhancement and the control of sports injury risks. In particular, the mid-season camp period loading is an important requirement to maintain the gains obtained in the pre-season training programs throughout the season. In this context, sports clubs prefer regions with different physical conditions (sea level, high altitude etc.) for the camp periods and allocate serious budgets for this periods.

Previous studies largely focused on effects of the pre-season camp period on psychological state and physical performance in soccer players. However, few studies in the current literature focused on the mid-season camp period. To the best of authors knowledge, sports injury anxiety and physical performance responses to the mid-season camp period loading in professional soccer players has not been very well discussed. Therefore the aim of this study is to investigate the effects of 3-week mid-season camp period loading on sports injury anxiety level and physical performances of professional male soccer players.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in study
* not have any musculoskeletal disease

Exclusion Criteria:

* using any drugs or supplements
* with a history of moderate to major injury within last 6 months
* having any systemic disease

Ages: 19 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Sports Injury Anxiety | Three week
  Sports injury anxiety level will be assessed by the Sports Injury Anxiety Scale. This scale is a valid and reliable scale used to determine the injury anxiety levels of athletes. The scale, adapted to Turkish, a 5-point Likert-type scale and consists of 13 questions in total. The minimum score that can be obtained from the scale is 19, and the maximum score is 95. A high score indicates high injury anxiety.

SECONDARY OUTCOMES:
Muscle strength | Three week
  Quadriceps femoris muscle strength will be assessed by the Lafayette manual muscle tester (Lafayette Instrument Company, Lafayette IN, USA). This device is a valid and reliable method that is frequently used in the assessment of muscle strength.Before the assessment, participants will be asked to sit unsupported on the treatment bed and keep the knee of the extremity to be measured at 90° flexion. During the assessment, participants will be asked to perform maximum isometric contraction for 3 seconds with the muscle in which the muscle strength will be evaluated against the resistance to be applied with a manual muscle tester. The assessments will be repeated three times with one-minute intervals for the dominant side, and the average of the measured values will be used for analysis.
Flexibility | Three week
  Flexibility will be assessed by the sit-and-reach test. The testing box will be fixed to the wall, and participants will be asked to sit with their knees extended and the soles of their feet against the testing box. Then, participants will be asked to slowly reach forward as far as possible along the top of the box and to hold the position for two seconds without bending their knees. The average of the two trials will be used for analysis.
Dynamic balance | Three week
  Dynamic balance will be assessed by the Y balance test. The test is a valid and reliable method that was developed as a version of the star excursion balance test. Before the assessment, three tape measures will be positioned at 135° between the anterior direction and the posterolateral/posteromedial directions. The measurement will be done for the dominant side three times and the average of the endpoints that the participants could reach will be used for data analysis. Reach distances will be normalized to limb length by calculating the maximized reach distance (in the percentage of maximized reach distance) using the formula (excursion distance/limb length) × 100 = percentage of maximized reach distance. The composite score will be calculated by taking the sum of three reach directions divided by three times the limb length then multiplied by 100. The mean value for the Y balance composite score will be used for analysis.
Single-leg jump | Three week
  Single-leg jump will be assessed by the single-leg jump test. The test is a valid and reliable method used in the assessment of jump performance in many studies. The participants will be asked to perform a single deep squat with a pause, followed by a vertical jump to maximum height with the dominant leg on the floor. This test will be performed three times for the dominant leg and the highest distance will be used for analysis.
Agility | Three week
  Agility will be assessed by the t-test. The t-test is a valid and reliable method used in the assessment of agility performance. For this test, an agility circuit will be created with four cones named 1, 2, 3, and 4. Cones will be placed at a distance of 9.14 m between 1 and 2, and 4.57 m between 2 and 3, and 2 and 4. At the "go" command, the participant will run forward as quickly as possible from cone 1 to cone 2, sidestepped to cone 3, sidestepped to cone 4, sidestepped to cone 2, then will run back as quickly as possible to cone 1. A stopwatch will be used during the test. All participants will perform the test 2 times with at least 2-minute rest periods between trials. The average of the two trials will be used for analysis.
Sprint | Three week
  Sprint performance will be assessed by the 20-m sprint test. The test is a valid and reliable method used in studies to assess sprint performance. During the test, at the "go" command, the participants will be asked to complete the 20-meter distance as quickly as possible, and a stopwatch will be used to determine the time to complete the test. All participants will perform the test two times with at least two minute rest periods between trials. The average of the two trials will be used for data analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Erhan Seçer, Manisa, Turkey (Türkiye)